CLINICAL TRIAL: NCT04839211
Title: Effects of High Intensity Interval-Based Inspiratory Muscle Training in Patients With Heart Failure
Brief Title: Inspiratory Muscle Training in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Dokuz Eylül University, Scientific Research Projects Coordination Unit (Unknown)
Responsible Party: Principal Investigator, Aylin Tanriverdi, Research assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3763-GOA
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): High-intensity interval-based inspiratory muscle training
  Interventions: Device: Inspiratory muscle training
- Sham inspiratory muscle training (Sham Comparator): Unloaded inspiratory muscle training
  Interventions: Device: Sham inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — Inspiratory muscle training will be performed three sessions per week as one supervised and two unsupervised for 8 weeks using an inspiratory muscle training device (PowerBreath). The inspiratory muscle training session will consist of 7 cycles including a 2:1 ratio of work and rest interval. Resistance will be adjusted to the highest tolerable load and will be gradually increased.
  Arms: Inspiratory muscle training
Device: Sham inspiratory muscle training — Sham inspiratory muscle training will be performed three sessions per week as one supervised and two unsupervised for 8 weeks using an inspiratory muscle training device (PowerBreath). The inspiratory muscle training session will consist of 7 cycles including a 2:1 ratio of work and rest interval. Resistance will be adjusted to the unloaded.
  Arms: Sham inspiratory muscle training

SUMMARY:
The aim of this study is to investigate the potential effects of inspiratory muscle training on cardiovascular, respiratory, physical, and psychosocial functions in patients with heart failure.

DETAILED DESCRIPTION:
Heart failure is a syndrome that leads to decreased cardiac output, inflammation, increased catabolism, and prolonged immobilization, causing inspiratory muscle weakness. Cardiac rehabilitation is a well-known treatment approach in heart failure however, the participation rate in cardiac rehabilitation is low. Therefore, inspiratory muscle training may serve as an alternative approach in patients with heart failure.

Patients will be randomly allocated into the inspiratory muscle training group and control group. The inspiratory muscle training (IMT) group will carry out IMT sessions three days per week for 8 weeks by using an inspiratory threshold loading device. Each session will consist of seven cycles including 2 min of breathing on an inspiratory loading device followed by 1 min of rest and will last 21 min. IMT will be performed at the tolerable maximum load for each 2-min work interval and will be progressively increased over the 8 weeks. The control group will perform unloaded IMT by using an inspiratory threshold loading device during all training sessions. Data will be collected before and after the treatment by a masked outcome assessor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with reduced ejection fraction
* Clinically stable
* Functional class II-III according to the New York Heart Association functional classification
* Having inspiratory muscle weakness (MIP<70%)
* Volunteer to participation

Exclusion Criteria:

* Congenital heart disease
* Severe valvular heart disease
* Cardiac device such as implantable cardioverter defibrillator or cardiac resynchronization therapy
* Neurological disease
* Conditions that may limit the physical mobility

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | change from baseline to 8 weeks
  Heart rate variability analysis, which gives information about the cardiac autonomic function, will be obtained from a short-term 5-min ECG recording using a SphygmoCor device.
Arterial stiffness | change from baseline to 8 weeks
  Arterial stiffness will be measured using a SphygmoCor device.

SECONDARY OUTCOMES:
Maximal inspiratory pressure | change from baseline to 8 weeks
  Maximal inspiratory pressure (MIP) will be measured using an electronic mouth pressure device. A higher inspiratory pressure indicates better inspiratory muscle strength.
Maximal expiratory pressure | change from baseline to 8 weeks
  Maximal expiratory pressure (MEP) will be measured using an electronic mouth pressure device. A higher expiratory pressure indicates better expiratory muscle strength.
Respiratory muscle endurance | change from baseline to 8 weeks
  Respiratory muscle endurance will be measured using an inspiratory muscle training device (PowerBreath). Higher values indicate better respiratory muscle endurance.
Forced vital capacity (FVC) | change from baseline to 8 weeks
  Forced vital capacity will be measured using a spirometer
Forced expiratory volume in 1 second (FEV1) | change from baseline to 8 weeks
  The pulmonary function will be measured using a spirometer
Forced expiratory flow at 25-75% of the vital capacity (FEF 25-75%) | change from baseline to 8 weeks
  Forced expiratory flow at 25-75% of the vital capacity will be measured using a spirometer
Dyspnea | change from baseline to 8 weeks
  Dyspnea will be assessed with the modified Medical Research Council (mMRC) scale.
  mMRC is a scale of 5 items (0-4). Higher scores indicate higher dyspnea perception.
Diaphragm thickness | change from baseline to 8 weeks
  Diaphragm thickness will be measured using a two-dimensional ultrasound machine.
Quadriceps muscle strength | change from baseline to 8 weeks
  Quadriceps muscle strength will be measured using a dynamometer. Higher values indicate better quadriceps muscle strength.
Balance | change from baseline to 8 weeks
  Balance performance will be assessed with a Balance Master System.
Functional capacity | change from baseline to 8 weeks
  Functional capacity will be assessed with 6 minute walk test.
Physical activity | change from baseline to 8 weeks
  Physical activity will be assessed with an activity monitor (SenseWear Armband) for consecutive 7 days.
Frailty | change from baseline to 8 weeks
  Physical frailty will be assessed with Field Frailty Phenotype. Field Frailty Phenotype consists of 5 criteria and scores 0 to 5. A score of 3-5 indicates frailty.
Fatigue | change from baseline to 8 weeks
  Fatigue will be assessed with Fatigue Impact Scale. Fatigue Impact Scale is a 40-item questionnaire. Each item is scored from 0-4 (a 4-point severity scale). The highest score is 160.
Disease-specific quality of life | change from baseline to 8 weeks
  Disease-specific quality of life will be assessed with Minnesota Living with Heart Failure Questionnaire. It is a 21-item questionnaire. Each item is scored from 0-5 (a 5-point severity scale). The highest score is 105.
Health-related quality of life | change from baseline to 8 weeks
  Health-related quality of life will be assessed with Short-Form 36 Health Survey Questionnaire (SF-36). SF-36 consists of 8 domains. Higher scores indicate a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Savci, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanriverdi A, Savci S, Ozcan Kahraman B, Odaman H, Ozpelit E, Senturk B, Ozsoy I, Baran A, Akdeniz B, Acar S, Balci A. Effects of high intensity interval-based inspiratory muscle training in patients with heart failure: A single-blind randomized controlled trial. Heart Lung. 2023 Nov-Dec;62:1-8. doi: 10.1016/j.hrtlng.2023.05.011. Epub 2023 Jun 7. PMID 37285766